CLINICAL TRIAL: NCT02459977
Title: The Usefulness of Tacrolimus Without Basiliximab in Well Matched Living Renal Transplantation in Korea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Su-Kil Park, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0209
Record Dates: First submitted 2015-04-28; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Basiliximab; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No basiliximab group (Experimental): The investigators omit basiliximab induction therapy in one to three-HLA mismatched living donor renal transplants.
  Interventions: Drug: No basiliximab; Procedure: Kidney transplantation
- Basilixiab group (Active Comparator): Age and sex matched patients who underwent one to three-HLA mismatched living donor renal transplants with basiliximab induction therapy (Control group)
  Interventions: Drug: Basiliximab; Procedure: Kidney transplantation

INTERVENTIONS:
Drug: Basiliximab — Basiliximab induction therapy
  Arms: Basilixiab group
Drug: No basiliximab — No basiliximab induction therapy
  Arms: No basiliximab group
Procedure: Kidney transplantation — kidney transplantation

SUMMARY:
Basiliximab has been a routine induction therapeutic agent even for well-matched living kidney transplantation(KT) with tacrolimus-based immunosuppression in Korea. As tacrolimus is a different drug from cyclosporine, the investigators study the usefulness of tacrolimus-based immunosuppression without basiliximab in well matched living KT.

DETAILED DESCRIPTION:
The investigators omit basiliximab induction therapy in patients who underwent one to three-HLA mismatched living donor renal transplantation. Participants should receive ABO compatible and T-flow negative transplants. The investigators compare the results of intervention group with conventionally treated control group (age and sex matched patient who underwent one to three-HLA mismatched living donor renal transplants with basiliximab induction therapy).

ELIGIBILITY:
Inclusion Criteria:

* ABO compatible and T-flow negative transplants
* Living kidney transplantation
* Tacrolimus based immunosuppression

Exclusion Criteria:

* Multiorgan transplantation
* Zero-mismatch transplantation (we use cyclosporine instead of FK506)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of rejection | within 3 years
  The investigators measures incidence of rejection by serum creatinine, urinalysis and kidney allograft biopsy.

SECONDARY OUTCOMES:
Incidence of infection | postoperative 6 month, 1 year, 1.5 year, 2 years and 3 years
  The investigators measures incidence of infection such as CMV, BKV infection, pneumonia, urinary tract infection and other infections.

CONTACTS AND LOCATIONS:
Overall Officials: Su-Kil Park, M.D, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea